CLINICAL TRIAL: NCT06071286
Title: SEQUENTIAL PROFILING OF TUMOR-DERIVED CIRCULATING CELL-FREE DNA (ctDNA) TO DETECT MINIMAL RESIDUAL DISEASE AND EARLY RELAPSE IN ADVANCED OVARIAN CANCER PATIENTS
Brief Title: SEQUENTIAL PROFILING OF TUMOR-DERIVED CIRCULATING CELL-FREE DNA (ctDNA) IN ADVANCED OVARIAN CANCER PATIENTS
Acronym: SPEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6065
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Patients with suspected advanced OC, based on preoperative imaging/clinical evaluation, will undergo blood samples in different timepoints
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — Patients with suspected advanced OC, based on preoperative imaging/clinical evaluation, will undergo blood samples in different timepoints

SUMMARY:
Ovarian cancer (OC) is the third most common gynaecologic cancer worldwide and has the highest mortality rate among gynaecologic cancers. Despite the advances in cytoreductive surgery and frontline chemotherapy, recurrence is a common event in the advanced disease setting, with more than 70% of women experiencing relapse within two years from diagnosis.

New strategies to anticipate the diagnosis of recurrence have been investigated in the last years. In this context, standard serum biomarkers, such as CA-125, and radiological evaluation are commonly used for disease surveillance, However, the early identification of relapsed disease as well as the identification of patients at higher risk for recurrence are still unmetclinical needs. Novel and reliable molecular biomarkers, which might also better represent the intrinsic molecular complexity of OC, could help clinicians to address this important challenge.

Circulating tumor DNA (ctDNA) analysis has recently emerged as a non-invasive tool to profile and monitor tumor evolution over time. CtDNA has been extensively studied in several neoplasms in order to evaluate its ability in anticipating detection of relapse compared to common markers used in clinical practice. Wehave designed a study to assess the ability of ctDNA to detect recurrence and progression of disease and to provide a genomic characterization, during follow-up of patients with advanced OC. If proven effective and reliable, ctDNA could be introduced into routine surveillance programme for OC.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed suspicious International Federation of Gynecology and Obstetrics (FIGO) stage III A or greater ovarian, fallopian tube, or primary peritoneal cancer
2. Age between 18 and 80 years
3. Estimated life expectancy of at least 4 weeks 4. Signed informed consent

Exclusion Criteria:

1. Any previous cancer in the last 5 years
2. Previous chemotherapy or target treatments 3. Diagnosis of synchronous tumors
3. Pregnancy or breastfeeding
4. Missed informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the ability of ctDNA to detect Ovarian Cancer recurrence. predictive value (NPV)). | 24 months
  The primary endpoint is to evaluate the ability of ctDNA to detect OC recurrence earlier than radiology (CT scan and ultrasound examination) and serum biomarkers used in clinical practice, in terms of diagnostic accuracy (i.e. specificity, sensitivity, positive predictive value (PPV) and negative predictive value (NPV)).

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Nero, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No